CLINICAL TRIAL: NCT03063775
Title: Proof of Concept: Intra-oral Soft Tissue Preservation of Extraction Sockets in Anterior Upper Jaw
Brief Title: Proof of Concept: Socket Seal
Acronym: SocketSeal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of suitable patients for recruitment
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7333
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Tissue Preservation
MeSH Terms: interventions — fibrinopeptides gamma; Bio-Oss; Fibrin Foam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 1. Mucograft® Seal + Bio-Oss® (Active Comparator)
  Interventions: Device: BioOss® + Mucograft Seal®
- 2. FGG + Bio-Oss® (Active Comparator)
  Interventions: Other: FGG + Bio-Oss®
- 3. FGG + Gelatine sponge (Spongostan®) (Active Comparator)
  Interventions: Other: FGG + Gelatine sponge (Spongostan®)
- 4. Spongostan®+ Mucograft® Seal (Active Comparator)
  Interventions: Device: Spongostan®+ Mucograft® Seal
- 5. Spongostan® (No Intervention)

INTERVENTIONS:
Device: BioOss® + Mucograft Seal® — Placement of BioOss®-Collagen into the extraction socket. The Mucograft Seal® Membrane is then applied to the socket.
  Arms: 1. Mucograft® Seal + Bio-Oss®
Other: FGG + Bio-Oss® — Placement of BioOss®-Collagen into the extraction socket. The FGG is then attached to the socket.
  Arms: 2. FGG + Bio-Oss®
Other: FGG + Gelatine sponge (Spongostan®) — Placement of a Gelatine sponge into the extraction socket, then attaching the FGG to the socket.
  Arms: 3. FGG + Gelatine sponge (Spongostan®)
Device: Spongostan®+ Mucograft® Seal — Placement of a Gelatine sponge into the extraction socket, then attaching the Mucograft® Seal Membrane to the socket
  Arms: 4. Spongostan®+ Mucograft® Seal

SUMMARY:
It is planned to evaluate if a porcine collagen matrix (Mucograft Seal) is offering comparable results to free gingival grafts (FGG) in post-extraction tissue preservation. If so, this would provide a substantial benefit to the patient as the second intervention on the palate and the subsequent morbidity of the donor site is omitted.

DETAILED DESCRIPTION:
In a proof of concept 5 groups are compared in preserving soft- and hard tissue after tooth extraction in the esthetic zone:

1. Mucograft® Seal + Bio-Oss®
2. Free Gingival Graft (FGG) + Bio-Oss®
3. Free Gingival Graft + Gelatine sponge (Spongostan®)
4. Spongostan®+ Mucograft® Seal
5. Spongostan®

Volumetric changes of hard and soft tissues are recorded , 2/4/8 weeks and 3/6/12 months after extraction.

ELIGIBILITY:
Inclusion Criteria:

• Planned extraction in the upper front or premolar region

Exclusion Criteria:

* General risk situation (antiresorptive therapy, antiangiogenic therapy, history of local radiation therapy, heavy coagulation disorder, relevant allergies, dysregulated Diabetes mellitus, malignant diseases)
* Acute gingivitis
* Deep pockets (>5.5mm)
* Apical periodontitis on neighboring teeth
* Heavy smoker (>10/d)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Soft tissue volume | 2 weeks
Soft tissue volume | 4 weeks
Soft tissue volume | 8 weeks

SECONDARY OUTCOMES:
Bone volume | 3 months
Bone volume | 6 months
Bone volume | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No